CLINICAL TRIAL: NCT02841540
Title: An Open-label, Multicenter Phase 1 Trial to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Splicing Modulator H3B-8800 for Subjects With Myelodysplastic Syndromes, Acute Myeloid Leukemia, and Chronic Myelomonocytic Leukemia
Brief Title: A Study of H3B-8800 (RVT-2001) in Participants With Lower Risk Myelodysplastic Syndromes
Acronym: Encore-MDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated after conducting an interim analysis of the available data where it became evident that the observed efficacy results were not in alignment with the initially set expectations.
Sponsor: Hemavant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H3B-8800-G000-101; 2016-001792-70 (EudraCT Number)
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic
Keywords: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; H3B-8800 (RVT-2001); Splicing Modulator; CMML; AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — H3B-8800

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- H3B-8800 (RVT-2001) Dose Escalation (Experimental): H3B-8800 Acute Myeloid Leukemia or High Risk Myelodysplastic Syndromes/ Low Risk Myelodysplastic Syndromes/ Chronic Myelomonocytic Leukemia.
  Interventions: Drug: H3B-8800 (RVT-2001)
- H3B-8800 (RVT-2001) MDS Expansion (Experimental): Transfusion-dependent, lower-risk MDS subjects (very-low to intermediate risk categorization per IPSS-R) with missense mutations in SF3B1.
  Interventions: Drug: H3B-8800 (RVT-2001)
- H3B-8800 (RVT-2001) Dose Optimization (Experimental): Transfusion-dependent, lower-risk MDS subjects (very-low to intermediate risk categorization per IPSS-R) with missense mutations in SF3B1, and who have not been exposed to HMA's or lenalidomide in a prior line of therapy.
  Interventions: Drug: H3B-8800 (RVT-2001)

INTERVENTIONS:
Drug: H3B-8800 (RVT-2001) — H3B-8800 (RVT-2001) orally at specified doses and schedules.

SUMMARY:
A Phase 1, an Open-label, Multicenter Phase 1 Trial to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Splicing Modulator H3B-8800 (RVT-2001) for Subjects With Myelodysplastic Syndromes, Acute Myeloid Leukemia, and Chronic Myelomonocytic Leukemia

DETAILED DESCRIPTION:
This study is a Phase 1, open-label, first-in-human (FIH) study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of H3B-8800 (RVT-2001) in subset of participants with Myelodysplastic Syndromes (MDS), Acute Myeloid Leukemia (AML), or Chronic Myelomonocytic Leukemia (CMML). The study consists of three parts, the dose escalation part (Part 1) exploring multiple once daily (QD) schedules and MDS Expansion part (Part 2) and Dose Optimization part (Part 3) exploring dosing schedules in lower-risk MDS.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of MDS, CMML, or AML.

   For the MDS Expansion cohort, participants must be lower-risk MDS, defined as low or intermediate-1 risk categorization per International Prognostic Scoring System (IPSS) criteria that carries a missense SF3B1 mutation.

   For the Dose Optimization cohort, participants must be transfusion-dependent, lower-risk MDS, defined as very-low to intermediate risk categorization per IPSS-R criteria that carries a missense SF3B1 mutation.
2. Participants must meet the following criteria relevant to their specific diagnosis:

   A. Participants with higher-risk MDS/CMML must be intolerant of hypomethylating agents (HMAs) or not have responded to 4 treatment cycles of decitabine or 6 treatment cycles of azacitidine, or must have progressed at any point after initiation of an HMA.

   B. For the Dose Escalation portion, participants with lower-risk MDS/CMML must be transfusion-dependent for red blood cells or platelets.

   For the MDS expansion cohort, lower risk MDS participants must be RBC transfusion dependent according to IWG 2006 criteria and must also have failed erythropoiesis stimulating agents (ESA) or have serum erythropoietin (EPO) levels greater than (>) 500 units per liter (U/L).

   C. For the Dose Optimization cohort, lower-risk MDS participants must be RBC transfusion-dependent at baseline defined as ≥3 RBC units (concentrates) in 16-weeks in at least 2 transfusion episodes prior to the first dose of H3B-8800 (RVT-2001) and must also have failed ESA or have serum EPO levels > 500 U/L. Any ESA use should be discontinued ≥6 weeks prior to enrollment.

   D. Participants with AML must either refuse or not be considered candidates for intensive induction chemotherapy using consensus criteria for defining such participants.

   E. Participants with CMML must have been treated with at least one prior therapy (hydroxyurea or a hypomethylating agent [HMA]).
3. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
4. For MDS expansion and Dose optimization cohorts - absolute neutrophil count (ANC) greater than or equal to (>=) 500/ microliter (mcL) (0.5*10^9/L).
5. For expansion and Dose optimization cohorts- platelet count >50,000/mcL (50*10^9/L).
6. For Dose-optimization cohort: No prior HMA or lenalidomide in participants with lower-risk MDS.
7. Adequate baseline organ function.

Exclusion Criteria:

1. Diagnosis of a core binding factor leukemia (t(8;21), t(16;16) or inv(16)). Diagnosis of acute promyelocytic leukemia (t(15;17))
2. Participants are deemed candidate for hematopoietic stem cell transplants at the time of enrollment (for AML participants only).
3. Known prior or current retinal or optic nerve disease (example, Retinitis Pigmentosa, diabetic retinopathy, optic neuritis) not stable for at least 6 months.
4. History of clinically significant, uncorrected vitamin B12 or folate deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLTs) | Escalation Cycle 1 (28 days)
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From the first dose of study drug until 30 days after final dose of study drug (up to approximately 50 months)
  The type and frequency of AEs and SAEs using CTCAE v4.03, as well as changes in clinical laboratory values, ECG parameters, ophthalmologic examinations, and vital sign measurements.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 Through the Last Measurable Point (AUC0-t) | Up to Cycle 6 Day 15 (each cycle length=28 days)
  Plasma samples for PK analyses will be collected at predetermined timepoint and analyzed
Maximum Observed Plasma Concentration (Cmax) | Up to Cycle 6 Day 15 (each cycle length=28 days)
  Plasma samples for PK analyses will be collected at predetermined timepoint and analyzed
Time of Maximum Observed Plasma Concentration (Tmax) | Up to Cycle 6 Day 15 (each cycle length=28 days)
  Plasma samples for PK analyses will be collected at predetermined timepoint and analyzed
Number of Participants who Achieve Red Blood Cell (RBC) Transfusion Independence | Up to approximately 50 months
Number of Participants with Hematologic Improvement | Up to approximately 50 months
Objective Response Rate (ORR) | Up to approximately 50 months
  ORR will be defined as the percentage of participants achieving a best overall response of partial remission (PR) or complete remission (CR) (PR + CR), from first dose date until disease progression/recurrence. CR includes CR with incomplete blood count recovery (CRi) in AML participants and marrow CR in MDS participants and optimal marrow response in CMML participants. Response will be assessed by the Investigator and the independent central review based on 2006 International Working Group (IWG) response criteria for MDS, 2003 IWG criteria for AML, and the international consortium proposal of uniform response criteria for CMML published in 2015.
Duration of Response (DOR) | Up to approximately 50 months
  DOR will be defined as the time from the date of first documented CR/PR until the first documentation of confirmed relapse, or death, whichever comes first.
Time to Progression | Up to approximately 50 months
Overall Survival (OS) | Up to approximately 50 months
  Overall Survival is defined as the time from first dose date to the date of death from any cause.
Mortality Rate at 3 and 6 Months | Months 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Keisuke Kuida, MD, PhD, Study Director — Hemavant Sciences
Locations (49):
- United States (15):
  - Arizona Oncology Associates, Tucson, Arizona
  - City of Hope, Duarte, California
  - City of Hope, Irvine, California
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Oncology Associates of Oregon, Eugene, Oregon
  - Texas Oncology, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialist, Fairfax, Virginia
- Belgium (4):
  - Algemeen Ziekenhuis Klina, Brasschaat
  - AZ Sint-Jan Brugge Oostende AV, Bruges
  - Universiteit Gent, Ghent
  - University Hospitals Leuven, Leuven
- France (7):
  - Institut Gustave Roussy, Villejuif, Val-de-Marne
  - CHU Amiens-Picardie, Amiens
  - Centre Hospitalier Universitaire d'Angers (CHU d'Angers), Angers
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Bordeaux
  - Centre Hospitalier - Le Mans, Le Mans
  - Hôpital Claude Huriez, Lille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Italy (4):
  - Azienda Ospedaliera Universitaria di Bologna - Policlinico S. Orsola Malpighi, Bologna
  - Fondazione IRCCS Cà Granda Ospedale Policlinico Maggiore, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - IRCCS Istituto Clinico Humanitas Cancer Center, Rozzano
- South Korea (8):
  - National Cancer Center, Gyeonggi-do, Goyang-si
  - Daegu Catholic University Medical Center, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
- Spain (6):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Valle de Hebrón, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario y Politécnico La Fe de Valencia, Valencia
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Chang-Gung Memorial Hospital, Chiayi, Chiayi City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Derived] Foran JM, Sanz GF, Watts JM, Brunner AM, Fossard G, Della Porta MG, Tsai XC, Garcia-Manero G, Dimicoli-Salazar S, Fletcher L, Kim YJ, Font P, Alfonso-Pierola A, Alonso-Dominguez JM, Benton C, Hong J, Malcovati L, Mazure D, Lee JH, Yeh SP, Goursaud L, Barcellini W, Wu E, Corzo D, Kuida K, Stone RM. Phase 1 first-in-human dose-expansion study of the oral SF3B1 modulator H3B-8800 in lower-risk myelodysplastic syndrome. Leuk Res. 2025 Sep;156:107735. doi: 10.1016/j.leukres.2025.107735. Epub 2025 Jun 9. PMID 40651101